CLINICAL TRIAL: NCT05322954
Title: Safety and Feasibility of Psilocybin in Methamphetamine Use Disorder in a Community-Based Sample
Brief Title: Study of the Safety and Feasibility of Psilocybin in Adults With Methamphetamine Use Disorder
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Revive Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-1087; 2021-1087 (Other: UW Madison); A532017 (Other: UW Madison); SMPH/FAMILYMEDICINE/FAMILYMED (Other: UW Madison); Protocol Version 7/11/2023 (Other: UW Madison)
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Use Disorder; Substance-Related Disorders; Chemically-Induced Disorders; Substance Use Disorders; Stimulant-Use Disorder
Keywords: methamphetamine; psilocybin; psychedelics; stimulants; substance use
MeSH Terms: conditions — Substance-Related Disorders; Chemically-Induced Disorders | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Psilocybin (Experimental): Psilocybin with psychological support: Psilocybin will be administered in the form of capsules, taken orally with water. Each participant will receive 2 doses, approximately 4 weeks apart.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 25mg orally followed by 25 mg or 50 mg orally

SUMMARY:
The purpose of this research study is to investigate the safety and feasibility of two (2) oral doses of psilocybin when combined with behavioral support for methamphetamine use disorder (MUD). Participants have a diagnosis of methamphetamine use disorder (MUD). Participants can expect to be actively engaged in the study for up to 26 weeks.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety of psilocybin in adult participants with MUD.

Eligible participants will be adults with methamphetamine use disorder recruited from the community. After physical and psychological screening, and at least 6 hours of psychological support for the psilocybin dosing, each participant will ingest 1 oral dose of psilocybin. All dosing sessions will be attended by 2 specially trained facilitators, in a dedicated Session Room at the University of Wisconsin School of Pharmacy. After eight hours of observation in the dosing room, the participant will stay overnight in the hospital Clinical Research Unit, and complete an integration session with at least one of the session facilitators before discharge to home. Approximately 4 weeks after the first dose, the participant will receive a second oral dose of psilocybin, with the same length of observation.

Participants who decide not to proceed to the second dose will complete two additional integration sessions and study measures through the two-month follow-up.

If you are interested in participating in this study, please fill out a brief 1-minute survey at the link in the "More Information" section at the bottom of this record.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of methamphetamine use disorder

Exclusion Criteria:

* Positive urine pregnancy at any time point during screening or study participation
* Inadequately treated hypertension, defined as 2 blood pressure readings, 10 minutes apart, of greater than 140/90 mmHg systolic/diastolic
* Current acute coronary syndrome or angina
* History of heart transplant or stroke
* Current use of and inability or unwillingness to taper off of medications that may interact with psilocybin
* Current insulin dependence, due to Type I or Type II diabetes

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events associated with oral psilocybin | Up to 26 weeks
  Incidence of serious adverse events attributable to psilocybin as categorized according to NCI Common Toxicity Criteria version 4.0. and assigned attribution (probably, possibly, and not related).

SECONDARY OUTCOMES:
Number of participants who complete at least one dose of psilocybin | Up to 26 weeks
  Study protocol retention and adherence for preparation, dosing and follow-up visits determined by adherence and retention rates, number of visits attended throughout the duration of the study.
Number of participants who complete two-month follow-up visit | Up to 26 weeks
  Study protocol adherence for preparation, dosing and follow-up visits determined by adherence and retention rates, number of visits attended throughout the duration of the study.
Changes in substance use | Up to 26 weeks
  Frequency of use of methamphetamine and other substances will be evaluated and tracked based on participant self-reported use at each visit.
Functional changes in psychedelic and addiction-related neurocircuitry using functional magnetic resonance imaging. | Up to 26 weeks
  Changes in functional connectivity (FC). Participants will undergo a 15-minute resting-state fMRI scanning sequence to measure changes in FC at rest pre- and post-dose.

OTHER OUTCOMES:
Changes in addiction-related constructs | Up to 26 weeks
  Changes in psychological, affective, and behavioral addiction-related constructs (e.g. craving, motivation, self-efficacy, self-compassion, mindfulness, experiential avoidance, etc.) measured by brief questionnaires prior to and following each psilocybin dosing session

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nicholas, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click this link to contact us to see if you qualify — https://redcap.ictr.wisc.edu/surveys/?s=7P8YKYW4EMWKCEHT